CLINICAL TRIAL: NCT04990180
Title: The Development and Feasibility Testing of a Pulmonary Rehabilitation Shared Decision Making Intervention for Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Pulmonary Rehabilitation Shared Decision Making Intervention
Acronym: PReSent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EDGE: 137907
Record Dates: First submitted 2021-07-14; First posted 2021-08-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Rehabilitation; Shared Decision Making; Patient Decision Aid; Decision Coaching; Implicit Association Test; Implicit Bias
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bias, Implicit

STUDY DESIGN:
Intervention Model Description: Mixed methods observational and feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shared Decision Making Intervention (Experimental): The intervention is a shared decision making consultation supported by a patient decision aid and decision coaching for healthcare professionals.
  Interventions: Behavioral: Shared Decision Making Intervention

INTERVENTIONS:
Behavioral: Shared Decision Making Intervention — Decision coaching will be provided to the Pulmonary Rehabilitation Specialists to provide the skills needed to facilitate shared decision making between themselves and patients (and carers). The patient decision aid will be an informational booklet which describes the available Pulmonary Rehabilitation options at the University Hospitals of Leicester. It will detail the risks and benefits of each option and provide interactive sections to engage patients with the content, guide them through it, encourage them to attribute personal meaning and preference to each one so they can make an informed and values-based decision about PR.

SUMMARY:
The PReSent study seeks to clarify the need, develop and test the feasibility and acceptability of a shared decision making intervention to support patients with Chronic Obstructive Pulmonary Disease make decisions about Pulmonary Rehabilitation. The study is split into two parts; (1) an observational study of healthcare professionals implicit attitudes, and (2) a feasibility and acceptability study assessing the value of the newly developed shared decision making intervention including a patient decision aid and decision coaching.

DETAILED DESCRIPTION:
Whilst Pulmonary Rehabilitation (PR) is an evidence-based intervention for patients with Chronic Obstructive Pulmonary Disease (COPD), the service suffers poor referral and uptake. One identified barrier to accessing PR at the University Hospitals of Leicester is healthcare professionals beliefs about patient motivation (e.g. believing patients to be unmotivated reduces their desire to offer PR). This shows healthcare professionals have conscious (explicit) bias but little is known about whether they also have unconscious (implicit) bias. It is important to measure this as it can also shape individuals attitudes and therefore referral behaviour.

The first objective of this study is to measure healthcare professionals implicit bias. Healthcare professionals from the United Kingdom who refer patients to PR will be invited to complete a one-off computerised Implicit Association Test, adapted to measure their bias towards the behaviours of patients living with COPD (i.e. smoking, exercising).

The second objective of this study is to test the feasibility and acceptability of a shared decision making intervention (a patient decision aid and decision coaching for PR specialists). Patients with COPD will receive the decision aid upon referral to PR and encouraged to use it to support their PR decision making. At their PR assessment they will engage in a shared decision making consultation with their trained PR specialist to decide on their preferred PR programme.

Following completion/drop out from PR, patients and trained PR specialists will be invited to take part in either a focus group (patients) or interview (PR specialist) to discuss the acceptability of the intervention.

ELIGIBILITY:
Phase 1: Measuring Healthcare Professionals attitudes towards patients with COPD

Inclusion Criteria:

* Willing and able to provide informed consent for participation in the research
* A United Kingdom healthcare professional
* A healthcare professional who has the capability to refer patients with COPD to Pulmonary Rehabilitation services
* Male or female, aged 18+ years
* Able to communicate in written and spoken English

Exclusion Criteria:

* Unable to provide valid informed consent
* Healthcare professionals practising outside of the United Kingdom
* A healthcare professional who does not refer patients with COPD to Pulmonary Rehabilitation services
* Aged <18 years
* Unable to understand written English as the Implicit Association Test is currently only available in English

Phase 2: A Pulmonary Rehabilitation shared decision making intervention Patients:-

Inclusion Criteria:

* Willing and able to give informed consent for participation in the research
* Male or female, aged 40+years
* A confirmed diagnosis of COPD, post bronchodilator Forced Expiratory Volume 1/Full Vital Capacity ratio <70%
* Eligible for attendance at a University Hospitals of Leicester Pulmonary Rehabilitation assessment
* Able to communicate in written and spoken English

Exclusion Criteria:

* Unable to provide valid informed consent
* Aged <40years
* Primary diagnosis is another chronic respiratory condition.
* Ineligible for attendance at a University Hospitals of Leicester PR assessment (e.g. significant comorbidity which limits exercise training
* Unable to understand written English as the research information and shared decision making intervention is currently only available in English

Healthcare professionals:-

Inclusion Criteria:

* A participant who is willing and able to give informed consent for participation in the research
* A healthcare professional directly involved in the provision of the shared decision making intervention (e.g. a Pulmonary Rehabilitation specialist)
* Male or female, aged 18+ years

Exclusion criteria:-

* A participant who is unable to provide valid informed consent
* A healthcare professional not directly involved in the provision of the shared decision making intervention
* Aged <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Response latency | Baseline only
  Presence of bias between stimuli
Feasibility of recruitment assessed by rate of recruitment to time and target | Through study completion, an average of 1 year
  Recruitment to time (proposed study end date) and target (proposed sample size)
Feasibility of data collection/outcome measures assessed by rate of participant attrition | 1 year (end of study)
  Data completeness
Intervention fidelity assessed by the Observer OPTION 5 Scale | 1 year (end of study)
  This questionnaire is completed by the researcher when listening back to the shared decision making consultation audio recordings. It measures adherence to the principles of shared decision making. It is a 5 item questionnaire with a 4 point Likert Scale with scores ranging from 0-20. The higher the score the greater the adherence to the principles of shared decision making.

SECONDARY OUTCOMES:
Decisional conflict measured using the Decisional Conflict Scale | Baseline & immediately post intervention
  The Decisional Conflict Scale is a self-reported, 16 item questionnaire with a 5 point Likert Scale with scores ranging from 0-64. The lower the score indicates lower decisional conflict.
Patient activation as measured by the Patient Activation Measure | Baseline & immediately post intervention
  The Patient Activation Measure is a self-reported, 13 item questionnaire with a 5 point Likert Scale. Raw scores are transformed to a scaled score between of 0-100 with 100 indicating the highest activation in self-management.
Rate of attendance assessed by the proportion of participants who complete the intervention | Baseline & immediately post intervention
  Intervention completion is termed as the number of participants who attend the shared decision making consultation.
Patient attitudes/experiences of the study assessed through qualitative interviews with study participants | 1 year (end of study)
  Patient attitudes/experiences of receiving the intervention
Health professionals attitudes/experiences assessed through qualitative interviews with study participants | 1 year (end of study)
  Health professional attitudes/experiences of delivering the intervention
Uptake and adherence to Pulmonary Rehabilitation assessed by the proportion of participants who begin and complete Pulmonary Rehabilitation | Baseline & immediately post intervention
  Completion is termed as participants who complete at least 8 of the available 12 sessions (75%).
COPD Assessment Test | Baseline & immediately post intervention
  The COPD Assessment Test is a self-reported, 8 item questionnaire with a 6 point Likert Scale with scores ranging from 0-40. Higher scores indicate lower health-related quality of life.
Bristol COPD Knowledge Questionnaire | Baseline & immediately post intervention
  The Bristol COPD Knowledge questionnaire is a multiple choice, 65 item self-reported questionnaire. Scores range from 0-65 with higher scores indicating greater knowledge of COPD.
Chronic Respiratory Questionnaire | Baseline & immediately post intervention
  The Chronic Respiratory Questionnaire is a self-reported 20 item questionnaire using a 7 point Likert Scale. Scores range from 7-140 with higher scores indicating greater health-related quality of life.
Hospital Anxiety and Depression Scale | Baseline & immediately post intervention
  The Hospital Anxiety and Depression Scale is a multiple choice, 14 item questionnaire using a 4 point Likert scale. Scores range from 0-42 with higher scores indicating greater levels of anxiety and/or depression.
COPD Prem 9 | Baseline & immediately post intervention
  The COPD Prem 9 is a self-reported, 9 item questionnaire with a 6 point Likert scale. Scores range from 0-45 with lower scores indicating better health-related quality of life.
Medical Research Council Dyspnoea Scale | Baseline & immediately post intervention
  The Medical Research Council Dyspnoea Scale is a self-reported, 1 item questionnaire using a 5 point Likert Scale. Scores range from 1-5 with higher scores indicating greater perceived breathlessness.
Incremental Shuttle Walking Test | Baseline & immediately post intervention
  Maximal exercise capacity test
Endurance Shuttle Walking Test | Baseline & immediately post intervention
  Maximal exercise capacity test
Patient satisfaction with Pulmonary Rehabilitation assessed by internal hospital satisfaction questionnaire | Baseline & immediately post intervention
  This is a 6 item open ended questionnaire exploring patient satisfaction with Pulmonary Rehabilitation. The text is analysed using qualitative research methods.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Direct access will be granted to authorised representatives from the Sponsor, host institution and the regulatory authorities to permit trial-related monitoring, audits and inspections- in line with participant consent.

REFERENCES:
- [Derived] Barradell AC, Doe G, Bekker HL, Houchen-Wolloff L, Robertson N, Singh SJ. A shared decision-making intervention for individuals living with chronic obstructive pulmonary disease who are considering the menu of pulmonary rehabilitation treatment options; a feasibility study. Chron Respir Dis. 2024 Jan-Dec;21:14799731241238428. doi: 10.1177/14799731241238428. PMID 39254860